CLINICAL TRIAL: NCT03862144
Title: One Day Antiemetic Prophylaxis of NEPA (Netupitant Plus Palonosetron) and Dexamethasone to Prevent Chemotherapy-induced Nausea and Vomiting (CINV) in Breast Cancer Patients Receiving an AC-based Chemotherapy Regimen
Brief Title: NEPA to Prevent Chemotherapy Induced Nausea and Vomiting in Patients With Breast Cancer
Acronym: GIM15-NEPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GIM15-NEPA
Record Dates: First submitted 2019-01-14; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: nausea; vomiting; breast cancer; AC-based chemotherapy
MeSH Terms: conditions — Vomiting; Nausea; Breast Neoplasms | interventions — netupitant, palosentron drug combination; netupitant; Palonosetron

STUDY DESIGN:
Intervention Model Description: Phase II study, one stage Fleming design, open-label, multicenter, not comparative
Oversight: Data Monitoring Committee: No

ARMS (1):
- Netupitant/Palonosetron & Dexamethasone (Experimental): * Netupitant/Palonosetron (NEPA) will be administered orally at the dose of 300 MG (milligrams) netupitant/0.5 palonosetron 1 hour before the start of any chemotherapy cycle.
  * Dexamethasone 12 mg will be added on day 1 only of each cycle.
  Interventions: Drug: Netupitant/Palonosetron

INTERVENTIONS:
Drug: Netupitant/Palonosetron
  Other Names: Netupitant/Palonosetron 300 MG-0.5 MG Oral Capsule [AKYNZEO]

SUMMARY:
This study evaluates if the activity of one-day of NEPA plus dexamethasone, to prevent chemotherapy-induced nausea and vomiting in breast cancer patients receiving adjuvant AC-based chemotherapy, is maintained during all the chemotherapy cycle treatment (maximum 4 cycles).

DETAILED DESCRIPTION:
Patients included in the study should be treated with the following antiemetic prophylaxis, during all the AC-based chemotherapy cycles, up to a maximum of 4 cycles:

* NEPA will be administered orally at the dose of 300 mg netupitant/0.5 palonosetron 1 hour before the start of any chemotherapy cycle.
* Dexamethasone 12 mg will be added on day 1 only of each cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years old
2. Histologically or cytologically confirmed diagnosis of breast cancer
3. Naïve patients
4. Be scheduled to receive adjuvant chemotherapy with anthracycline (doxorubicin or epirubicin) + cyclophosphamide (AC-based regimen)
5. ECOG (Eastern Cooperative Oncology Group) performance status 0-2
6. Body Mass index (BMI) ≥ 18.5
7. Written informed consent
8. If women of childbearing potential age: reliable contraceptive measures must be used during the study treatment period and up to 30 days after last NEPA administration
9. Acceptable hepatic function (<= 2 times the upper limit of normal for liver transaminases) and renal function (creatinine < 1.5 times the upper limit of normal);
10. Ability and willingness of the patient to complete the diary.

Exclusion Criteria:

1. Advanced/metastatic breast cancer
2. Patients already submitted to non-AC-based chemotherapy
3. Treatment with investigational medications in 30 days before NEPA
4. Myocardial infarction within the last 6 months
5. Documented or known hypersensitivity to 5HT3RA (5-Hydroxytryptamine Receptor 3 Antagonists) or NK1RA (Neurokinin-1 Receptor Antagonists) and excipients
6. Uncontrolled diabetes mellitus
7. Nausea and vomiting at baseline
8. Chronic use of other antiemetic agent(s)
9. Patient's inability to take oral medication
10. Gastrointestinal obstruction or active peptic ulcer
11. Pregnancy or breastfeeding
12. Prior malignancies at other sites except surgically treated non-melanoma skin cancer, superficial cervical cancer, or other cancer from which the patient had been disease-free for ≥ 5 years
13. Psychiatric or CNS (Central Nervous System) disorders interfering with ability to comply with study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
Complete response | During the overall phase (From day 1 to day 5 after any AC-based chemotherapy administration) for a maximum 4 cycles (each cycle is 21 days)
  The rate of patients achieving and maintaining a complete response (defined as no emetic episode and no use of rescue medication) during the overall phase of all AC-based chemotherapy cycles

SECONDARY OUTCOMES:
Acute and Delayed Phase Complete Response | During the Acute Phase [0-24 hours after chemotherapy (CT)] and the Delayed (25-120 hours) phase
  Rate of complete control (defined as no emetic episode and no need for rescue medication)
Complete Control | During the Acute Phase (0-24 hours after chemotherapy), the Delayed (25-120 hours), the Overall (0-120 hours) phases for each cycle and separately on single days of all chemotherapy cycles (each cycle is 21 days), up to 4 cycles
  Rate of complete control (defined as complete response with a maximum grade of mild nausea)
Emesis-Free | During the Acute (0-24 hours after CT), the Delayed (25-120 hours), the Overall (0-120 hours) phases for each cycle (each cycle is 21 days)and separately on single days of all CT cycles,up to 4 cycles.Also during the period between two consecutive cycles
  Percentage of emesis-free patients (no emetic episodes) after any AC-based chemotherapy administration.
Nausea | During the Acute (0-24 hours after CT), the Delayed (25-120 hours), the Overall (0-120 hours) phases for each cycle (of 21 days)and separately on single days of all chemotherapy cycles, up to 4 cycles.Also during the period between two consecutive cycles
  Presence of nausea graded according to Likert scale (none, mild, moderate and severe)
Global satisfaction with antiemetic therapy: Visual Analogue Scale (VAS) | During the Acute Phase (0-24 hours after CT), the Delayed (25-120 hours), the Overall (0-120 hours) phases for each cycle (each cycle is 21 days) and separately on single days of all CT cycles, up to 4 cycles
  Patient global satisfaction with antiemetic therapy, as measured by a Visual Analogue Scale (VAS). Scale ranges are 0-10 (0 represents maximum dissatisfaction, 10 represents maximum satisfaction)
Safety profile (according to CTCAE) | During the Acute Phase (0-24 hours after CT), the Delayed (25-120 hours), the Overall (0-120 hours) phases for each cycle (each cycle is 21 days) and separately on single days of all CT cycles, up to 4 cycles
  Safety profile according to CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Michelino De Laurentiis, MD, PhD, Principal Investigator — National Cancer Institute "Fondazione Pascale", Naples

REFERENCES:
- [Derived] Caputo R, Cazzaniga ME, Sbrana A, Torrisi R, Paris I, Giordano M, Montesarchio V, Guarneri V, Amaducci L, Bilancia D, Cilenti G, Fabi A, Collova E, Schirone A, Bonizzoni E, Celio L, De Placido S, De Laurentiis M. Netupitant/palonosetron (NEPA) and dexamethasone for prevention of emesis in breast cancer patients receiving adjuvant anthracycline plus cyclophosphamide: a multi-cycle, phase II study. BMC Cancer. 2020 Mar 19;20(1):232. doi: 10.1186/s12885-020-6707-9. PMID 32188417